CLINICAL TRIAL: NCT00658866
Title: Target Site Pharmacokinetics of Ertapenem After Multiple Doses in Diabetes Patients With Soft Tissue Infection
Acronym: 2007-005020-33
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Markus Mueller, Medical University of Vienna, Department of Clinical Pharmacology
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Erta_MD_1
Record Dates: First submitted 2008-04-04; First posted 2008-04-15 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-03

CONDITIONS: Soft Tissue Infection
Keywords: ertapenem tissue PK
MeSH Terms: conditions — Soft Tissue Infections | interventions — Microdialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Microdialysis — PK measurements with microdialysis

SUMMARY:
Background/rationale: Ertapenem is an innovative antimicrobial agent, which is approved in the European Union for diabetic foot infections of the skin and soft tissue. Although its antimicrobial spectrum and activity against ESBL-strains are promising to treat infected ulcers associated with diabetes, there is a lack of data on tissue pharmacokinetics of ertapenem in this patient population. However, for antimicrobial efficacy it is important to show that the antibiotic achieves sufficient concentrations at the site of infection, i.e. in tissue. A recent clinical study by Burkhardt et al. (Journal of Antimicrobial Chemotherapy, 2006) using the microdialysis technique showed that the free tissue concentrations after a single dose of 1 g ertapenem are sufficient and adequate to kill most relevant bacteria, suggesting efficacy of ertapenem for soft tissue infections. It is well known that there is no accumulation of ertapenem in plasma after multiple doses of 1 g every 24 h in patients without significantly impaired renal function. The single dose study by Burkhardt et al. also suggests that only negligible drug accumulation can be expected in soft tissues of healthy young volunteers after multiple doses. However, it was shown for other antibiotics that tissue PK may be significantly different under pathologic conditions, leading to impaired penetration, but subsequent accumulation after multiple doses due to a longer tissue half life than in healthy volunteers. Since the properties of inflamed tissue may diverge from those of healthy tissue it is important to evaluate which concentrations of ertapenem are reached in inflamed tissue after multiple doses.

Clinical study: In the present study we will measure the concentrations of ertapenem over time in plasma and infected tissue of 10 diabetes patients after multiple doses. The microdialysis technique will be used. The ertapenem concentrations will be measured in inflamed tissue and in non-inflamed subcutaneous tissue to identify the effect of inflammation on pharmacokinetics. The findings of the present study will help to confirm the efficacy of ertapenem for the indication of diabetic soft tissue infections.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 18 and 85 years
* Diagnosis of Diabetes mellitus
* Clinically diagnosed skin or soft tissue infection and/or infected ulcers of the leg, requiring antimicrobial therapy
* Prescription of ertapenem for therapeutic reasons
* Willingness and ability to comply with the protocol
* Signed informed consent

Exclusion Criteria:

* HIV, Hepatitis B or C positive
* Allergy or hypersensitivity against study drug
* Severe renal impairment, defined by a serum creatinine level > 1.6 mg/L
* Pregnancy, or women of child bearing potential not willing to apply adequate contraception during study period
* Any disease considered relevant for proper performance of the study, or risks to the patient, at the discretion of the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics in tissue | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Markus Mueller, MD, Principal Investigator — Medical University of Vienna, Dep. of Clinical Pharmacology
Locations (1):
- Medical University Vienna, Department of Clinical Pharacology, Vienna, Vienna, Austria